CLINICAL TRIAL: NCT07403123
Title: Competitive Swimmer, Swimmer's Shoulder, Forward Head Posture, Round Shoulder Posture
Brief Title: The Effect of Exercise Intervention on Forward Head Posture and Round Shoulder Posture in Symptomatic Competitive Swimmer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Fu-Jie Kang, Assistant professor, Fooyin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKU HREC-E-112-082-2
Record Dates: First submitted 2026-01-20; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Swimmer Shoulder; Forward Head Posture; Posture and Mobility of the Upper Quadrant
Keywords: swimmer shoulder; forward head posture; round shoulder posture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group performed an exercise program targeting RSP and FHP, which included three strengthening exercises and two stretching exercises. Each session lasted approximately 50 minutes and was conducted three times per week for a total of eight weeks.
  Interventions: Other: exercise intervention: included three strengthening exercises and two stretching exercises.
- non-intervention group (No Intervention): The non-intervention group did not receive the above exercise training during the eight-week intervention period; however, the relevant exercise training was provided after the completion of the eight-week experiment.

INTERVENTIONS:
Other: exercise intervention: included three strengthening exercises and two stretching exercises. — Strengthening exercises: Based on the relevant literature review, the primary aim of the strengthening exercises was to enhance the strength of the middle trapezius, lower trapezius, and serratus anterior muscles, including: Y to W exercise, L to Y exercise and Scapular protraction exercise.
  Stretching exercises: Based on a review of the relevant literature, stretching exercises primarily target the pectoralis minor and the cervical extensor muscles, including: Pectoralis flexibility and Chin tucks exercise.
  Arms: intervention group

SUMMARY:
This study is an exercise intervention study, and its findings will help to clarify the effects of exercise on forward head posture and rounded shoulder posture in competitive swimmers. It is expected that the results of this study will assist in ensuring that forward head posture and rounded shoulder posture are taken into consideration when competitive swimmers undergo related exercise training in the future. The purpose of this experiment is purely for academic research and does not constitute a physical examination or a medical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. High school competitive swimmers
2. With shoulder pain: unilateral or bilateral shoulder pain who had a self-reported shoulder pain score of ≥ 40 points for at least one month, measured using a visual analogue scale (VAS). VAS scores range from 0 to 100, with higher scores indicating greater pain.
3. With round shoulder posture (RSP): Forward shoulder angle (FSA) ≥ 52°.
4. With forward head posture (FHP): forward head angle (FHA) ≥ 46°.

Exclusion Criteria:

1. A history of fractures
2. Previous surgery to the upper extremity or shoulder joint
3. Full-thickness rotator cuff tears
4. Cervical radiculopathy
5. Shoulder dislocation
6. Structural deformities of the cervical or thoracic spine
7. Any neurological disorder

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
forward head angle (FHA) | Both groups underwent baseline posture assessments prior to the intervention and post-intervention posture assessments at the end of the 8-week training period.
  The forward head angle (FHA) (Degree): The FHA is defined as the angle formed by the intersection of two lines: one vertical line passing through the spinous process of the seventh cervical vertebra (C7), and a second line connecting the C7 spinous process to the tragus of the ear. A larger FHA value indicates a more severe FHP. The examiner photographed the standing posture. The photograph was then analyzed using AutoCAD software (AutoDesk Inc., Sausalito, CA) to calculate the FHA (forward head angle) value.
forward shoulder angle (FSA) | Both groups underwent baseline posture assessments prior to the intervention and post-intervention posture assessments at the end of the 8-week training period.
  The FSA (forward shoulder angle) (Degree): The FSA is defined as the angle formed by the intersection of two lines: one vertical line passing through the spinous process of the seventh cervical vertebra (C7), and a second line connecting the C7 spinous process to the center of the humerus. A larger FSA value indicates a more severe RSP. The examiner photographed the standing posture. The photograph was then analyzed using AutoCAD software (AutoDesk Inc., Sausalito, CA) to calculate the FSA (forward shoulder angle) value.

SECONDARY OUTCOMES:
Pectoralis minor index (PMI) | Both groups underwent baseline assessments prior to the intervention and post-intervention assessments at the end of the 8-week training period.
  PMI (cm/cm): The examiner used a digital caliper to measure the distance between the inferomedial border of the coracoid process and the fourth rib-sternal junction. This measured distance (cm) was then divided by the participant's height (cm) and multiplied by 100 to obtain the PMI.
Shoulder pain and disability index (SPADI) | Both groups underwent baseline assessments prior to the intervention and post-intervention assessments at the end of the 8-week training period.
  SPADI: Shoulder pain and disability index (SPADI) was selected for assessment of shoulder pain and disability. Score from 0 to 10. Higher scores indicate greater pain and disability.
Scapular upward rotation (SUR) angle | Both groups underwent baseline assessments prior to the intervention and post-intervention assessments at the end of the 8-week training period.
  SUR (degree): Measurements were obtained using an ACUMAR™ digital inclinometer. Measurements were taken in three positions: with the arms resting at the sides, with the arms elevated to 60°, and with the arms elevated to 120° . SUR (°) was defined as the angle between the scapular spine and the horizontal reference line.
Scapular anterior tilt index (SATI) | Both groups underwent baseline assessments prior to the intervention and post-intervention assessments at the end of the 8-week training period.
  SATI: The participant lay supine on a bed in a relaxed position. The distance (cm) between the posterior border of the acromion and the bed surface was measured, and this value was then divided by 100 to obtain the SATI.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of physical therapy, Fooyin university, Kaohsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol